CLINICAL TRIAL: NCT06810856
Title: A Modified Draize Repeat Insult Patch Test in Healthy Volunteers, of Either Sex, to Investigate the Irritation and Allergenic Potential of One Test Article Following Repeated Cutaneous Patch Applications
Brief Title: HRIPT Study to Evaluate the Irritation and Allergenic Potential of Medical-grade Norway Spruce (Picea Abies) Resin Salve (Abilar)
Acronym: HRIPT-REPRIP2M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Repolar Pharmaceuticals Oy (Industry)
Collaborators: Princeton Consumer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REPRIP2M
Record Dates: First submitted 2025-01-24; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Skin Irritation; Skin Sensitization
Keywords: HRIPT; Skin Irritation; Contact Sensitization; Patch Testing; Dermatological Safety

STUDY DESIGN:
Intervention Model Description: This is a single-group interventional study in which all participants received the same topical test product applied via occlusive patches. The study was designed to evaluate skin irritation and sensitization potential using a repeat insult patch test protocol.
Masking Description: This study was conducted as a single-blind HRIPT, where participants were not informed of the identity of the test article applied to their skin. However, as only one test product was used without a control or comparison group, ClinicalTrials.gov does not allow classification as "Single-Blind," and the study is categorized as "Open Label" in this registration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical-Grade Norway Spruce Resin product (Abilar) Topical Safety Study (Experimental): Participants received repeated applications of a Medical-Grade Norway Spruce Resin product (Abilar) topical formulation using Finn chambers on Scanpor® tape. Patches were applied to the upper back for 47 hours per application over a three-week induction phase, followed by a challenge phase to assess potential delayed hypersensitivity reactions. Skin reactions were assessed at scheduled intervals by a blinded dermatologist using a standardized scoring system.
  Interventions: Device: Abilar® Resin Salve

INTERVENTIONS:
Device: Abilar® Resin Salve — Abilar® Resin Salve is a medical-grade Norway spruce (Picea abies) resin-based topical medical device, classified as a Class IIb medical device in the EU. It is designed for wound care and skin protection, forming a moist healing barrier while exhibiting antimicrobial properties. It contains 10% of medical-grade Picea abies resin.
  Other Names: Abilar; Abilar® 10% Resin Salve; Norway Spruce Resin-Based Topical Medical Device; Picea abies Resin Salve; Abilar Wound Salve

SUMMARY:
The goal of this clinical trial is to assess whether a medical-grade Norway spruce resin-based topical product (Abilar) causes skin irritation or allergic sensitization in healthy adult volunteers. The main questions it aims to answer are:

Does the product cause skin irritation after repeated applications? Does the product induce sensitization (allergic contact dermatitis) after repeated exposure?

Participants will:

Have the test product applied to their skin via occlusive patches multiple times over three weeks.

Undergo dermatological assessments for signs of erythema (redness), swelling, or sensitization at scheduled time points.

Have a final challenge application on a new skin site after a rest period to check for delayed allergic reactions.

This study follows Good Clinical Practice (GCP) guidelines and the Declaration of Helsinki. It was conducted at Princeton Consumer Research (PCR Corp, UK) with approval from the East Anglia Ethics Committee, UK.

DETAILED DESCRIPTION:
Study Objective:

This is a single-center, interventional study designed to evaluate the irritation and sensitization potential of a medical-grade Norway spruce resin-based wound care product (Abilar) using a Modified Draize Human Repeat Insult Patch Test (HRIPT). The study followed Good Clinical Practice (ICH GCP 1996) and the Declaration of Helsinki.

Study Design:

A total of 215 healthy adult volunteers were enrolled, with 207 completing the study. The study was conducted at Princeton Consumer Research (PCR Corp, UK) and was approved by the East Anglia Ethics Committee, UK. Participants received occlusive patches containing the test product, applied repeatedly over a three-week induction phase. After a rest period, a challenge application was placed on a new skin site to evaluate potential delayed-type hypersensitivity reactions.

Single-center, interventional study with single-group assignment (no control group).

Conducted under dermatological supervision at Princeton Consumer Research (PCR Corp, UK).

Ethical approval was granted by the East Anglia Ethics Committee, UK. Study Period: October 16, 2019 - October 25, 2019.

Methodology:

Induction Phase (Days 1-21): Repeated application of occlusive patches with the test product to the same skin site three times per week. Skin assessments were conducted at multiple time points.

Rest Period: No patch application for approximately 14 days. Challenge Phase (Day 38): A final application was made to a naïve skin site to assess delayed hypersensitivity responses.

Scoring System: Skin reactions were graded using dermatological visual scoring for erythema, edema, and other signs of irritation or sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, of either sex, aged at least 18 years.
* Completed written informed consent.

Exclusion Criteria:

* Pregnancy or lactation.
* Inadequate or non-existent contraception (women of child bearing potential only).
* A current skin disease of any type apart from mild facial acne (e.g. eczema, psoriasis).
* Heavy alcohol consumption (i.e. more than 21 units per week or 8 units a day for men, more than 14 units per week or 4 units a day for women).
* Current use or history of repeated use of street drugs.
* A febrile illness lasting more than 24 hours in the six days prior to first patch application.
* Significant past medical history of hepatic, renal, cardiac, pulmonary, digestive, haematological, neurological, locomotor or psychiatric disease.
* History of asthma only if requiring regular medication or hay fever that required prescription treatment in two or more of the previous three years.
* A history of multiple drug hypersensitivity.
* Concurrent medication likely to affect the response to the test articles or confuse the results of the study.
* Known sensitivity to the test articles or their constituents including patch materials.
* Current treatment by a physician for allergy unless physician consulted by Investigator and participation approved.
* Participation in a repeat insult patch test (RIPT) or follow-up work within the last month.
* Sensitisation or questionable sensitisation in a RIPT.
* Recent immunisation (less than 10 days prior to test patch application).
* A medical history indicating atopy.

Prohibitions and Restrictions:

* No use of aspirin or non-steroidal anti-inflammatory drugs for the duration of the study.
* No use of sun beds or sun lamps and no deliberate exposure of the test sites to natural sunlight for the duration of the study.
* No immunisation from ten days prior to first patching until study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Skin Irritation During Induction Phase | Days 1 to 22 (Induction Phase)
  The primary outcome measure was the percentage of participants exhibiting skin irritation reactions (e.g., erythema, edema, papules) at any time during the Induction Phase of the HRIPT study. Reactions were graded using a standardized visual scoring system.

SECONDARY OUTCOMES:
Incidence of Sensitization Reactions During Challenge Phase | Days 36 to 40 (Challenge Phase)
  This study assessed the presence of delayed hypersensitivity reactions following re-exposure to the test product after a rest period. Participants were evaluated one hour and 49 hours post-challenge patch removal using a standardized dermatological scoring system.

CONTACTS AND LOCATIONS:
Locations (1):
- Princeton Consumer Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected throughout the study, including anonymized participant-level skin reaction assessments, will be made available upon request for research purposes.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available upon request after study completion and final publication, with an access period of 5 years post-publication.
Access Criteria: Researchers requesting access to anonymized IPD must submit a written request outlining the intended research objectives. Data access will be granted following review and approval by the sponsor (Repolar Pharmaceuticals Oy) and compliance with data protection regulations.

REFERENCES:
- [Background] Jordan WP Jr, King SE. Delayed hypersensitivity in females. The development of allergic contact dermatitis in females during the comparison of two predictive patch tests. Contact Dermatitis. 1977 Feb;3(1):19-26. doi: 10.1111/j.1600-0536.1977.tb03582.x. PMID 844299
- See also: Related Info — https://www.repolar.com